CLINICAL TRIAL: NCT04541134
Title: A Multi-center, Randomized, Placebo-controlled, Double-blind, Cross-over, Phase 3 Clinical Trial to Evaluate of the Efficacy and Safety of DW9801 in Patients With Primary Dysmenorrhea
Brief Title: Phase 3 Clinical Trial to Evaluate of the Efficacy and Safety of DW9801 in Patients With Primary Dysmenorrhea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DW9801-303
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — pelubiprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other)
  Interventions: Drug: Pelubiprofen 45mg; Drug: Placebo
- Group 2 (Other)
  Interventions: Drug: Pelubiprofen 45mg; Drug: Placebo

INTERVENTIONS:
Drug: Pelubiprofen 45mg — Pelubiprofen 45mg 1 tab for moderate or severe menstrual pain, bid for 3days(prn)
Drug: Placebo — Placebo1 tab for moderate or severe menstrual pain, bid for 3days(prn)

SUMMARY:
A Multi-center, Randomized, Placebo-controlled, Double-blind, Cross-over, Phase 3 Clinical Trial to Evaluate of the Efficacy and Safety of DW9801 in Patients with Primary Dysmenorrhea

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age between 19 years to 44years
* Patients with menstrual pain over 4 out of 6 menstrual cycles before screening
* Patients with moderate or severe menstrual pain for recent 2 menstrual cycles
* Patients with regular menstrual cycles(28±7 days) for a year

Exclusion Criteria:

* Patients diagnosed or suspected of secondary dysmenorrhea
* Previous adverse reaction or known allergy to NSAIDs
* Breast feeding woman
* Patients who are not willing to use proper contraception during clinical trial period

Ages: 19 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
TOTPAR-8 | Day 1
  Time weighted sum of total pain relief
SPID-8 | Day 1
  Sum of pain intensity difference

IPD SHARING:
Plan to Share IPD: No